CLINICAL TRIAL: NCT02846246
Title: The Effects and Meaning of a Person-centred and Health-promoting Intervention in Home Care Services: Study Protocol of a Non-randomised Controlled Trial
Brief Title: The Effects and Meaning of a Person-centred and Health-promoting Intervention in Home Care Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, David Edvardsson, Professor, Umeå University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016/04-31Ö
Record Dates: First submitted 2016-07-12; First posted 2016-07-27 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Staff and Older Persons With Home Care Service
Keywords: aged care; health; home care services; person-centred care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The experimental group will be introduced to a person-centred care model that involves shared decision making where the person with home care service and family together with contact nurse prioritise care content and make rearrangements to make sure the provided home care service maximises health.
  Interventions: Other: Person-centred and health-promoting home care service
- Control (Sham Comparator): A usual care paradigm will guide the control units, i.e. a continuation with practice as usual.
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Person-centred and health-promoting home care service — Firstly, staff will take part in an educational program on the content and operationalization of the central theoretical components person-centeredness and health exploratory conversation. Secondly, staff will participate in supervised skill training in how to accomplish person-centered and health exploratory conversation. Thirdly, the staff will have a person-centred and health exploratory conversation with purpose to evaluate the extent to which current home care service practice meet the older person´s need and maintain or make rearrangement in provided care to maximise older people's health. Finally, staff will participate in clinical supervisory sessions with an aim to support and facilitate ongoing operationalization phase.
  Arms: Intervention
Other: Care as usual — The control group will be offered a lecture about dementia based on staff wishes and a usual care paradigm will guide the control units, i.e. a continuation with practice as usual. Control units will receive the intervention protocol and study results at the end of the study.
  Arms: Control

SUMMARY:
Current home care service are to a large extent task oriented with a limited focus on care recipient's involvement. Furthermore, studies have shown that low care recipients' involvement might decrease older people's quality of life. Person-centred care focusing on involvement has improved the quality of life and the satisfaction with care for older people in health care and nursing homes but there is a lack of knowledge about the effects and meaning of a person-centred interventions in aged care at home. Present study describes the evaluation of a person-centred and health-promoting intervention.

DETAILED DESCRIPTION:
This is a non-randomised controlled trial with a before-after approach. The investigators will include 270 home care recipients >65 years, 270 family members and 65 staff in intervention group and control group respectively. Participants will be recruited from a municipality in northern Sweden. The intervention involves letting the person and family together with contact nurse prioritise care content and make rearrangements to make sure the home care service maximises the potential to satisfy psychosocial, physical, and functional needs and increasing health. Outcome assessment will focus on; a) quality of life (primary outcomes), thriving and satisfaction with care for older people, b) caregiver strain, informal caregiving engagement and satisfaction with care for relatives, c) job satisfaction and stress for care staff. Evaluation will be performed by questionnaires and interviews.

Person-centred home care services have the potential to improve the recurrently reported sub-standard experiences of home care services and the study result will hopefully lead the way in establish a person-centred and health-promoting model in aged care and living conditions for older people.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for care recipients will be:

* persons 65 years or older
* living at home with granted HCS
* have at least two visits per month, and
* be Swedish speaking

Inclusion for family members:

* be defined by the care recipients as his/her family member, and
* Swedish speaking

Inclusion for staff:

* have an employment for more than 6 month in the HCS district at baseline, be a contact staff and
* Swedish speaking
* Care recipients who apply for HCS in the district during the study period will be offered the intervention but not be included in the evaluation

Exclusion Criteria

* No exclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change of Quality of Life assessed with the Nottingham Health Profile scale | Baseline, 12 and 24 month follow-up
  The Nottingham Health Profile scale will be used to assess quality of life. Nottingham health profile includes 38 items in six dimensions: energy level, pain, emotional reaction, sleep, social isolation, and physical abilities. Each item is answered through Yes/No statements and range from best (0) to worst (100) possible score. The Nottingham Health Profile has been found to be sensitive for changes, valid and reliable.
Change of Quality of Life assessed with the EQ-5D | Baseline, 12 and 24 month follow-up
  As a complement, the EQ-5D will also be used to assess quality of life. The EQ-5D consists of two parts, a health state description and a visual analogue scale. The health state description comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels on a Likert-scale: none (0) to extreme (4). The visual analogue scale rates participants overall health between endpoints, worst imaginable health (0) and best imaginable health (100). EQ-5D has been found to be sensitive for changes and valid.

SECONDARY OUTCOMES:
Change in thriving assessed with the Thriving of Older People Assessment Scale | baseline, 12 and 24 month follow-up
  Thriving will be assessed with The Thriving of Older People Assessment Scale which includes 32 items and consists of five sub-scales: resident attitude towards the place where they are living, quality of the care and care-givers, activities and peer relationships, opportunities to keep in touch with people and places of importance, and qualities in the physical environment. Each item has six answer alternatives on a Likert-scale ranging from No (1) to Yes, I agree completely (6). The Thriving of Older People Assessment Scale has been found to be valid and reliable.
Change in satisfaction with home care service assessed with the Quality of Care from the Patients' Perspective | baseline, 12 and 24 month follow-up
  Satisfaction with home care service will be measured with The Quality of Care from the Patients' Perspective which includes 64 items and consists of four dimensions: medical-technical competence (11 items), physical-technical conditions (10 items), identity-oriented approach (30 items) and social-cultural atmosphere (13 items). Each item should be answered in two ways; perceived reality and subjective importance. Perceived reality range between Not applicable (1) to Fully agree (5) on a five level Likert-scale while the subjective importance range between Of very great importance (1) to of little importance (4). The Quality of Care from the Patients' Perspective has been found to be valid and reliable.

OTHER OUTCOMES:
Change in informal caregiver strain assessed with the Caregiver Burden Scale | baseline, 12 and 24 month follow-up
  To assess informal caregiver strain, The Caregiver Burden Scale will be used. The scale includes 22 items in five dimensions: general strain, isolation, disappointment, emotional involvement, and environments. Response alternatives is a four-point Likert-scale: Not at all (1) to Often (4). The Caregiver Burden Scale has been found to be valid and reliable.
Change in informal caregiving engagement assessed with the Resource Utilization in Dementia instrument | baseline, 12 and 24 month follow-up
  Informal caregiver engagement will be assessed with The Resource Utilization in Dementia instrument which include three parts: personal activities of daily living (dressing/undressing, showering/bathing, washing, and moving), instrumental activities of daily living (cooking, shopping, washing, cleaning, taking care of economy, talking on the telephone, riding/driving car, and other transportations), and supervision (risks as fire, accidents, fall in house or outside etc.). The Resource Utilization in Dementia assesses resource utilization in terms of: hours of home care, number of days in hospital, number of visits to GP´s, physiotherapists, and informal care. The instrument has been found to be valid and reliable
Change in satisfaction with care for relatives assessed with the Pyramid questionnaire | baseline, 12 and 24 month follow-up
  Satisfaction with care will be assessed with The Pyramid questionnaire which includes 40 items in seven parts; information, staff professional skills, care, activity, contact, social support and relative participation. Response alternatives is a four-point Likert-scale: Yes, to a great degree to No, not at all. The scale has been found to be valid and reliable.
Change in job satisfaction assessed with the Measure of Job Satisfaction | baseline, 12 and 24 month follow-up
  Job satisfaction will be assessed with The Measure of Job Satisfaction which includes 37 items in five dimensions; personal satisfaction, satisfaction with workload, team spirit, training and professional support. Response alternatives is a five-point Likert-scale: Very dissatisfied (1) to Very Satisfied (5). The scale has been found to be valid and reliable.
Change in stress of conscience assessed with the Stress of Conscience scale | baseline, 12 and 24 month follow-up
  To assess stress of conscience, The Stress of Conscience scale will be used. the scale consists of ten items related to different health care situations, each question consists of an A and B part. The A parts' response alternatives are a six-point Likert-scale ranging from Never (0) to Every day (5). The questions are related to how often different situations arise at the workplace. The B parts are a ten centimetre visual analogue scale where each situations' impact on conscience are estimated. A total index can be calculated where a higher value means higher levels of stress of conscience. The Stress of Conscience scale has been found to be valid. A weakness is the absence of reliability test

CONTACTS AND LOCATIONS:
Overall Officials: David Edvardsson, Professor, Principal Investigator — Umea University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamas K, Bolenius K, Sandman PO, Lindkvist M, Edvardsson D. Effects of a person-centred and health-promoting intervention in home care services- a non-randomized controlled trial. BMC Geriatr. 2021 Dec 18;21(1):720. doi: 10.1186/s12877-021-02661-5. PMID 34922494
- [Derived] Bolenius K, Lamas K, Sandman PO, Lindkvist M, Edvardsson D. Perceptions of self-determination and quality of life among Swedish home care recipients - a cross-sectional study. BMC Geriatr. 2019 May 24;19(1):142. doi: 10.1186/s12877-019-1145-8. PMID 31126243
- [Derived] Bolenius K, Lamas K, Sandman PO, Edvardsson D. Effects and meanings of a person-centred and health-promoting intervention in home care services - a study protocol of a non-randomised controlled trial. BMC Geriatr. 2017 Feb 16;17(1):57. doi: 10.1186/s12877-017-0445-0. PMID 28209122